CLINICAL TRIAL: NCT04957602
Title: Evaluation of a Novel Microfluidic Device to Purify Metastatic Lung Cancer Patients CTC (Circulating Tumoral Cells and Enable Their Culture (in Vitro and in Ovo)
Brief Title: Evaluation of a Novel Microfluidic Device to Purify Metastatic Lung Cancer Patients CTC (Circulating Tumoral Cells)
Acronym: LUTON
Status: Terminated | Type: Observational
Why Stopped: funding ending
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0928; 2021-A01838-33 (Other: ID-RCB)
Record Dates: First submitted 2021-07-06; First posted 2021-07-12 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Non Small Cell Lung Cancer
Keywords: metastatic; non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic non-small cell lung cancer patients: Metastatic non-small cell lung cancer patients who have not initiated their treatment yet (osermertinib or chemotherapy (associated or not with immunotherapy)
  Interventions: Other: Blood collection

INTERVENTIONS:
Other: Blood collection — Blood collection (4*10ml) before treatment initiation and after the first evaluation (usually 3-4 months after treatment initiation).

SUMMARY:
Currents strategies for cancer diagnosis consist of the extraction of a solid tissue from the affected area. This sample enables the study of specific biomarkers and the genetic nature of the tumor.

However, the tissue extraction is risky and painful for the patient and in some cases is unavailable in inaccessible tumors.

In addition, cancer is a dynamic disease and during the course of disease, cancers generally become more heterogeneous. As a result of this heterogeneity, the bulk tumour might include a diverse collection of cells harbouring distinct molecular signatures with differential levels of sensitivity to treatment. This heterogeneity might result in a non-uniform distribution of genetically distinct tumour-cell subpopulations across and within disease sites (spatial heterogeneity) or temporal variations in the molecular makeup of cancer cells (temporal heterogeneity).

To overcome these drawbacks, new alternatives are rising up, such as liquid biopsy.

A liquid biopsy is the analysis of biomarkers in a non-solid biological tissue, mainly blood, which has remarkable advantages over the traditional method; it has no risk, it is non-invasive and painless, it does not require surgery and reduces cost and diagnosis time.

Of the various circulating biomarkers, circulating tumor cells (CTCs) have particularly opened new windows. Circulating tumor cells (CTCs) are released into the bloodstream from primary cancer, metastasis, and even from a disseminated tumor cell reservoir.

CTCs may ideally replace tissue biopsies in the prediction and monitoring of therapeutic responses and tumor recurrence. CTCs can be used to guide therapeutic cancer management and serve as drug targets.

There are a wide range of instruments and methods for capturing, enriching, and enumerating CTCs. However, none of them is considered optimal.

To improve the purity of CTCs, the study consortium has developed a cutting-edge microfluidic device (LUTON) to reduce leukocytes contamination while preserving CTCs viability.

The added-value of the study innovation has been validated on clinical cell lines. The aim of this study is now to determine the performance of the device using patients' blood samples.

For this purpose, CTCs from non-small cell lung metastatic cancer patients will be isolated using ClearCellFX1 before injection into the LUTON workflow.

Collected cells will then be either growth in vitro or in ovo and the added value of this extra step of purification determined.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patient (>18 years)
* Stage IV non-small cell lung cancer (depending on classification)
* First line treatment approved by Multidisciplinary Team Meeting (MDTM) and referent physician
* Able to provide non-objection to participation

Exclusion Criteria:

* Patient weight below 50kg at inclusion
* Suspected Pregnancy

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic non-small cell lung cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
2 days CTCs viability evaluation after purification by our innovative LUTON microfluidic device | 2 days after injection in the microfluidic device.
  Circulating Tumoral Cells (CTCs) from blood samples will be retrieved and enriched by ClearCellFX1 before being injected in the LUTON workflow. Purified CTCs will then be collected after their passage into the microfluidic device to be cultivate in 3D.
  After 2 Days, a "Live and Dead" test will be realized to quantified the amount of living cells (30 samples from diagnosis).

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien COURAUD, PhD, Principal Investigator — Service de Pneumologie Aiguë Spécialisée et Cancérologie thoracique
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France